CLINICAL TRIAL: NCT07387055
Title: The Effect of Artificial Intelligence on the Development of Projective Methods Used in the Determination of Dental Anxiety in Children
Brief Title: Effect of Artificial Intelligence on Assessing Dental Anxiety in Children
Status: Completed | Type: Observational
Sponsor: Sümeyra Akkoç (Other)
Responsible Party: Sponsor-Investigator, Sümeyra Akkoç, Assistant Professor, DDS, Kutahya Health Sciences University
Organization: Kutahya Health Sciences University (Other)
Other Study IDs: 2024/05-33
Record Dates: First submitted 2026-01-20; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Dental Anxiety; Artificial Intelligence (AI); Test Anxiety Scale
Keywords: Dental Anxiety; Pediatric Dentistry; Artificial Intelligence; Child-Dntist Interaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First Dental Visit Group: Children aged 3-6 years who presented for a routine dental examination, were attending their first dental visit, and met the inclusion and exclusion criteria constituted the study group.

SUMMARY:
The goal of this observational study was to evaluate an artificial intelligence-assisted projective method for assessing dental anxiety in young children and to understand how the first child-dentist interaction affected dental anxiety. The main questions it aimed to answer were:

Did the artificial intelligence-assisted projective method provide a valid and reliable assessment of dental anxiety in children aged 3 to 6 years? Did dental anxiety change after the child's first interaction with the dentist during the first dental visit? Children aged 3 to 6 years who attended their first dental visit as part of routine dental care took part. During the same visit, dental anxiety was assessed before and after the initial child-dentist interaction using picture-based dental anxiety scales and the newly developed projective method. All assessments were completed on the same day.

DETAILED DESCRIPTION:
This study evaluated the validity and reliability of an artificial intelligence-assisted projective assessment tool using the Facial Image Scale, the Venham Picture Test, and the Raghavendra, Madhuri, and Sujata Pictorial Scale as comparator measures. Dental anxiety was assessed with the AI-assisted tool and all comparator scales immediately before and immediately after the child's first interaction with the dentist during the same visit. Reliability was evaluated using the intraclass correlation coefficient (ICC), agreement was assessed using Bland-Altman analysis, and criterion validity was assessed using Spearman rank correlation. Pre-interaction and post-interaction dental anxiety scores were compared using the Wilcoxon signed-rank test separately for each measurement tool.

ELIGIBILITY:
Inclusion Criteria:

* The child and the parent/guardian agree to participate in the study.
* The child's native language is Turkish.
* The child is attending their first dental visit.
* The child has no systemic disease.
* The child is able to cooperate sufficiently to complete the initial dental examination.

Exclusion Criteria:

* Current use of medication, a known history of allergy, or the presence of any mental or physical disability

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 3-6 years who presented for a routine dental examination to the Department of Pediatric Dentistry, Kütahya Health Sciences University, between August 2024 and November 2024.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
AI-Assisted Projective Dental Anxiety Assessment Tool Score | Immediately before and immediately after the initial child-dentist interaction (same visit)
  Dental anxiety is assessed using an AI-Assisted projective assessment tool. The score ranges from 1 to 5, and higher scores indicate higher dental anxiety.
Facial Image Scale (FIS) Score | Immediately before and immediately after the initial child-dentist interaction (same visit)
  Dental anxiety is assessed using the FIS. The score ranges from 1 to 5, and higher scores indicate higher dental anxiety.
Venham Picture Test (VPT) Score | Immediately before and immediately after the initial child-dentist interaction (same visit)
  Dental anxiety is assessed using the VPT. The score ranges from 0 to 8, and higher scores indicate higher dental anxiety.
Raghavendra, Madhuri, and Sujata Pictorial Scale (RMS-PS) Score | Immediately before and immediately after the initial child-dentist interaction (same visit)
  Dental anxiety is assessed using the RMS-PS. The score ranges from 1 to 5, and higher scores indicate higher dental anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Kütahya Health Sciences University, Faculty of Dentistry, Department of Pediatric Dentistry, Kütahya, Centre, Turkey (Türkiye)